CLINICAL TRIAL: NCT06144996
Title: Development of a Canadian Bronchiectasis and NTM Database
Status: Recruiting | Type: Observational
Sponsor: University of Calgary (Other)
Collaborators: Insmed Incorporated (Industry); Trudell Medical International (Industry)
Responsible Party: Sponsor
Other Study IDs: REB21-1131
Record Dates: First submitted 2023-06-28; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-06

CONDITIONS: Bronchiectasis; Non-Tuberculous Mycobacterial Pneumonia
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-CF Bronchiectasis Patients with or without NTM: Patients over the age of 18 with non-CF Bronchiectasis with or without Nontuberculosis Mycobacteria (NTM).
- Nontuberculosis Mycobacteria (NTM): Patients over the age of 18 with Nontuberculosis Mycobacteria (NTM)

SUMMARY:
The investigators aim to develop a comprehensive patient registry of patients with non-CF bronchiectasis and/or Nontuberculosis Mycobacteria (NTM)

DETAILED DESCRIPTION:
The investigators aim to develop a comprehensive patient registry of patients with non-CF bronchiectasis and/or Nontuberculosis Mycobacteria (NTM). This will entail inclusion of adults (age >18 years) with a diagnosis of these conditions to be entered with complete clinical data and quality of life assessments entered into a patient registry.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18
* Non-CF Bronchiectasis
* Nontuberculosis Mycobacteria (NTM)

Exclusion Criteria:

* Under the age of 18
* CF bronchiectasis

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18 with non-CF Bronchiectasis and/or Nontuberculosis Mycobacteria (NTM).
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2050-01 (Estimated); Study Completion 2050-01 (Estimated)

PRIMARY OUTCOMES:
Patient Recruitment and Data analysis for NTM and Bronchiectasis | December 2050
  Descriptive analysis of demographics and clinical parameters and epidemiological evaluation of No. of hospitalizations, No. of exacerbations.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No